CLINICAL TRIAL: NCT06348225
Title: Post-exercise Hot Water Immersion to Improve Blood Pressure Control
Brief Title: Post-exercise Hot Water Immersion to Improve Overnight Blood Pressure
Acronym: ExHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Providence College (Other)
Responsible Party: Principal Investigator, Brett Romano Ely, Assistant Professor of Health Sciences, Providence College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FY24-10
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Elevated Blood Pressure
Keywords: exercise, heat therapy
MeSH Terms: conditions — Hypertension; Motor Activity; Hyperthermia | interventions — Exercise; Diathermy

STUDY DESIGN:
Intervention Model Description: A repeated-measures design will be used with all participants completing the three acute interventions (exercise, heat, or exercise + heat) as well as a control day.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask the participant to treatments (exercise/no exercise, water temperature, etc) or the PI who is monitoring them during treatment. However, all data (hourly blood pressure, heart rate variability, and flow-mediated dilation) will be analyzed by an individual blinded to the trial/intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise + Heat Therapy (Experimental): This treatment will include exercise (treadmill walking) and hot leg bath.
  Interventions: Behavioral: Exercise; Other: Heat Therapy
- Heat Therapy (Experimental): This treatment will only include the hot leg bath (no exercise).
  Interventions: Other: Heat Therapy
- Exercise (Active Comparator): This treatment will include exercise (treadmill walking) followed by a sham leg bath.
  Interventions: Behavioral: Exercise; Other: Sham leg bath
- Control (No Intervention): Participants will refrain from exercise or heat exposure for at least 24 hours, and perform all study analyses for a control comparison.

INTERVENTIONS:
Behavioral: Exercise — Participants will walk on a treadmill for 30 minutes at 55-60% of heart rate reserve. The treadmill will be set at 2mph and 2% grade, then be adjusted in the first 5 minutes to achieve target heart rate.
  Other Names: Treadmill walking
  Arms: Exercise; Exercise + Heat Therapy
Other: Heat Therapy — Participants will place their legs in a deep leg bath (mid-calf) set to 42C for 45 minutes.
  Other Names: hot leg bath
  Arms: Exercise + Heat Therapy; Heat Therapy
Other: Sham leg bath — Participants will place their legs in a deep leg bath (mid-calf) set to 36C for 45 minutes.
  Other Names: lukewarm leg bath
  Arms: Exercise

SUMMARY:
The goal of this clinical trial is to test whether putting a participant's legs in a hot bath after exercise improves blood pressure in people with higher blood pressure.

. The main questions it aims to answer are:

* Whether exercise alone, hot water leg bath alone, or both treatments together cause blood pressure to be lower during sleep.
* If there are any changes in heart rhythm or blood vessel health after exercise, hot water leg bath, or the two treatments together that relate to changes in blood pressure.

Participants will complete four different trials:

* 30 minutes of walking with a 45-minute lukewarm leg bath after
* 30 minutes of walking with a 45-minute hot leg bath after
* 45 minutes of a hot leg bath with no exercise
* A day with no exercise or leg bath Researchers will look at heart rhythm, blood vessels, and blood pressure after each of these trials to see if there are differences, and if exercise and heat together can improve heart health more than exercise or heat alone.

DETAILED DESCRIPTION:
In 2017, the American Heart Association updated standards for diagnosing hypertension, while emphasizing the need for lifestyle modification in the early stages of blood pressure elevation. Using these updated criteria, approximately 1/3 of U.S. adults have hypertension, but few are able to improve blood pressure through diet and exercise and often progress to more severe disease states. Novel interventions to promote blood pressure reduction in mild hypertension are needed to attenuate or prevent this progression to more severe hypertension. Heat therapy, the repeated application of passive heat through hot water immersion, has gained recent attention for promising blood pressure reduction and improvement in cardiovascular health. Preliminary work combining exercise and hot water leg immersion indicates improved overnight blood pressure in individuals with elevated blood pressure, but the magnitude and mechanisms of this improvement require further study.

It is unknown whether the decrease in blood pressure following post-exercise heat exposure results from changes in systemic regulation (autonomic nervous system function, measured through heart rate variability), local factors (improved blood vessel function, measured through flow-mediated dilation), or both. The goal of the proposed research is to examine the impact of exercise alone (30 minutes of treadmill walking), hot water immersion alone (45 minutes in a leg bath set to 42°C), and combined exercise + hot water immersion (30 minutes treadmill walking followed by 45 minutes in a 42°C leg bath) on nocturnal blood pressure, autonomic function, and blood vessel function in individuals with elevated blood pressure. This goal will be addressed with the following specific aims:

Aim 1. To examine the impact of exercise, hot water leg immersion, or combined exercise + hot water immersion on overnight blood pressure in individuals with elevated blood pressure. The researchers hypothesize that the combination of exercise and hot water immersion will result in reduced systolic and diastolic blood pressure through 12 hours post-exercise as compared to baseline or either standalone treatment.

Aim 2. To examine changes in autonomic function, as measured by heart rate variability (HRV) following exercise, leg heating, or combined therapies. The researchers hypothesize that combined exercise and hot water immersion will result in higher HRV (indicating improved autonomic balance) compared to baseline measures.

Aim 3. To examine changes in blood vessel (endothelial) function, measured using flow-mediated dilation, following exercise, leg heating, or combined therapies. The researchers hypothesize that combined exercise and hot water immersion will result in a higher flow-mediated dilation (indicating improved blood vessel relaxation) compared to baseline or either standalone intervention.

The results of this study have important health implications in the treatment of hypertension using lifestyle interventions for the millions of Americans with elevated blood pressure or hypertension. The findings have the potential to improve non-pharmacological treatment of hypertension by developing an exercise and heat exposure protocol that is cost-effective, easily implemented, and results in substantially reduced blood pressure and improved cardiovascular risk profile.

ELIGIBILITY:
Inclusion Criteria:

* resting blood pressure >120/80 mmHg; measured at screening visit
* BMI between 18-39.9
* capable of walking 30 min at a moderate intensity on a treadmill

Exclusion Criteria:

* diagnosed hypertension
* taking antihypertensive medications
* history of heat injury or heat illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ambulatory blood pressure | 24 hours post-treatment
  Welch-Allyn ambulatory blood pressure monitor placed on the arm after treatment
Heart Rate Variability | 30-60 min post-treatment
  3-lead ECG with paced breathing measured post-treatment
Flow-mediated dilation | 30-60 min post-treatment
  Measure of endothelial function in the brachial artery (arm), change in blood vessel diameter following a 5-minute blood flow occlusion and release

CONTACTS AND LOCATIONS:
Overall Officials: Brett R Ely, PhD, Principal Investigator — Providence College
Locations (1):
- Providence College, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
The current plan is to share only compiled data with other researchers if requested.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT06348225/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT06348225/ICF_001.pdf